CLINICAL TRIAL: NCT02669914
Title: A Phase II Study of MEDI4736 (Durvalumab) in Patients With Brain Metastasis From Epithelial-derived Tumors
Brief Title: MEDI4736 (Durvalumab) in Patients With Brain Metastasis From Epithelial-derived Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual, funding withdrawn by AstraZeneca, and change in clinical practice
Sponsor: Washington University School of Medicine (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201602169
Record Dates: First submitted 2016-01-22; First posted 2016-02-01 (Estimated); Results first posted 2018-10-10 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-10

CONDITIONS: Non-Small Cell Lung Cancer; Nonsmall Cell Lung Cancer; Breast Cancer; Cancer of Breast; Cancer of the Breast; Gastroesophageal Cancer; Pancreatic Cancer; Cancer of the Pancreas; Colorectal Cancer; Colorectal Carcinoma; Renal Cancer; Kidney Cancer; Cancer of the Kidney; Cancer of Kidney; Ovarian Cancer; Ovary Cancer; Cancer of the Ovary; Cancer of Ovary
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Breast Neoplasms; Pancreatic Neoplasms; Colorectal Neoplasms; Kidney Neoplasms; Ovarian Neoplasms | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A: Non-small cell lung cancer w/o corticosteroids (Experimental): -MEDI4736 will be given to all patients > 30 kg actual body weight intravenously at a fixed dose 750 mg every 2 weeks over the course of 60 minutes on an outpatient basis on Days 1 and 15 of each 28-day cycle. Patients < 30 kg actual body weight will be dosed at 10 mg/kg every 2 weeks.
  Interventions: Drug: MEDI4736
- Cohort B: Epithelial origin solid tumors w/o corticosteroids (Experimental): -MEDI4736 will be given to all patients > 30 kg actual body weight intravenously at a fixed dose 750 mg every 2 weeks over the course of 60 minutes on an outpatient basis on Days 1 and 15 of each 28-day cycle. Patients < 30 kg actual body weight will be dosed at 10 mg/kg every 2 weeks.
  Interventions: Drug: MEDI4736
- Cohort C: NSCLC or non-NSCLC w/corticosteroids (Experimental): -MEDI4736 will be given to all patients > 30 kg actual body weight intravenously at a fixed dose 750 mg every 2 weeks over the course of 60 minutes on an outpatient basis on Days 1 and 15 of each 28-day cycle. Patients < 30 kg actual body weight will be dosed at 10 mg/kg every 2 weeks.
  Interventions: Drug: MEDI4736

INTERVENTIONS:
Drug: MEDI4736
  Other Names: Durvalumab

SUMMARY:
Brain metastases are the most common intracranial malignancy occurring in 20-40% of all cancers, and the presence of CNS metastases is associated with a poor prognosis. As such, the median overall survival of patients with symptomatic brain lesions is a dismal 2-3 months regardless of tumor type. Because standard chemotherapy largely does not cross the blood brain barrier at a meaningful concentration, standard treatment is limited and usually involves surgical resection and/or stereotactic radiosurgery for isolated lesions and whole brain radiation for multiple lesions. Unfortunately, the median overall survival is only improved by about 6 months with this multimodality approach2, and there is a paucity of second-line therapies to treat recurrence. Furthermore, re-resection and re-radiation are often not feasible options due to concern for increasing complications or neurotoxicity, respectively. Thus, there is a dire clinical need for additional treatment options for this patient population.

Checkpoint blockade therapy, in particular PD-1 and PD-L1 inhibition, has recently shown clinical efficacy in multiple types of solid tumors. The investigators propose to study the efficacy of checkpoint blockade therapy in patients with solid tumors and refractory/recurrent brain metastases. The investigators will assess the efficacy of MEDI4736, a novel PD-L1 inhibitory monoclonal antibody, in this study.

ELIGIBILITY:
Inclusion Criteria:

* Cohort A: Histologically confirmed metastatic non-small cell lung cancer (all histologic subtypes allowed) with radiographic evidence by MRI of at least one measurable brain lesion as defined by RANO criteria that does not require corticosteroids for symptomatic control.
* Cohort B: Histologically confirmed metastatic solid tumor of epithelial origin, excluding NSCLC, including but not limited to ovarian cancer, colorectal cancer, pancreatic cancer, gastric cancer, renal cancer, bladder cancer, or breast cancer with radiographic evidence by MRI of at least one measurable brain lesion as defined by RANO criteria that does not require corticosteroids for symptomatic control.
* Cohort C: Histologically confirmed metastatic solid tumor of epithelial origin, including both NSCLC and non-NSCLC, with radiographic evidence by MRI of at least one measurable brain lesion as defined by RANO criteria that requires corticosteroids for symptomatic control.
* At least one prior treatment to a CNS-based lesion is required. Prior therapy must be completed > 2 weeks prior to enrollment. A previously treated lesion must be demonstrated by MRI to have progressed following treatment in order to be eligible. The subsequent development of a new CNS lesion that was not previously treated will be permitted and dose not require treatment followed by progression prior to enrollment. Treatment of a single CNS lesion with local therapy in the context of multifocal disease is permitted as long as at least one untreated lesions meets criteria for measurable disease. Patients should have received minimum of one line of systemic therapy.
* At least 18 years of age.
* ECOG performance status of 0 to 2
* Adequate bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelets ≥ 100,000/mcL
  * Hemoglobin ≥ 8.0 g/dL
  * Serum bilirubin ≤ 1.5 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 x IULN
  * Creatinine clearance ≥ 40 mL/min/1.73 m2 by the Cockcroft-Gault formula or by 24-hour urine collection for determination of creatinine clearance
* Negative antiviral serology:

  * Negative human immunodeficiency virus (HIV) antibody.
  * Negative hepatitis B surface antigen (HBsAg) and negative hepatitis B core (HBc) antibody or undetectable hepatitis B (HBV) DNA by quantitative polymerase chain reaction (PCR) testing.
  * Negative hepatitis C virus (HCV) antibody or negative HCV ribonucleic acid (RNA) by quantitative PCR.
* Mean QT interval corrected for heart rate (QTc) < 470 msec calculated from 3 ECGs performed at least 2 minutes apart using Frediricia's Correction.
* Female subjects must either be of non-reproductive potential (i.e., post-menopausal by history: ≥60 years old and no menses for 1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Diagnosis of leptomeningeal carcinomatosis.
* Diagnosis of melanoma or other non-epithelial based malignancy such as sarcoma, neuroendocrine tumor, small cell lung cancer.
* Presence of unstable systemic disease (e.g., visceral crisis or rapid progression) in the judgment of the investigator.
* A history of other malignancy ≤ 5 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only or carcinoma in situ of the cervix.
* Currently receiving any other investigational agents.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to MEDI4736 or other agents used in the study.
* Previous treatment with a PD-1 or PD-L1 inhibitor, including MEDI4736, or a CTLA-4 inhibitory agent.
* Current or prior use of immunosuppressive medication within 28 days before the first dose of MEDI4736 with the exceptions of intranasal and inhaled corticosteroids, or systemic corticosteroids in Cohort C.
* Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) 21 days prior to the first dose of study drug.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension (>180/110), unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses, or psychiatric illness/social situations that would limit compliance with study requirements.
* Active or prior documented autoimmune disease within the past 2 years (Note: subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded).
* Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
* History of prior immunodeficiency.
* History of allogeneic organ transplant.
* Known history of previous clinical diagnosis of tuberculosis.
* Receipt of live attenuated vaccination within 30 days prior to first dose of MEDI4736.
* Pregnant and/or breastfeeding or female patients of reproductive potential who are not employing an effective method of birth control.
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-09-12 (Actual); Primary Completion 2017-09-21 (Actual); Study Completion 2018-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramaswamy Govindan, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 09/12/2016 and closed to participant accrual on 11/16/2017.
Period: Overall Study
Arm/Group | Cohort A: Non-small Cell Lung Cancer w/o Corticosteroids | Cohort B: Epithelial Origin Solid Tumors w/o Corticosteroids | Cohort C: NSCLC or Non-NSCLC w/Corticosteroids
Started | 4 | 0 | 0
Completed | 4 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: There were not any participants enrolled in Cohort B or Cohort C so that is why the overall number of baseline participants is zero for these cohorts.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Non-small Cell Lung Cancer w/o Corticosteroids | Cohort B: Epithelial Origin Solid Tumors w/o Corticosteroids | Cohort C: NSCLC or Non-NSCLC w/Corticosteroids | Total
Number analyzed (Participants) | 4 | 0 | 0 | 4
Age, Continuous [Median (Full Range); unit: years] | 62 [55 to 76] |  |  | 62 [55 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 |  |  | 3
  Male | 1 |  |  | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  |  | 0
  Not Hispanic or Latino | 4 |  |  | 4
  Unknown or Not Reported | 0 |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  | 0
  Asian | 0 |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  |  | 0
  Black or African American | 1 |  |  | 1
  White | 3 |  |  | 3
  More than one race | 0 |  |  | 0
  Unknown or Not Reported | 0 |  |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 |  |  | 4

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate of Intracranial Disease
Description: -% of subjects who achieve a complete response (CR) or partial response (CR) based on assessment of brain lesions
  * CR: Requires: complete disappearance of all enhancing measurable and nonmeasurable disease sustained for at least 4 weeks; No new lesions; stable or improved nonenhancing (T2/FLAIR) lesions.; off corticosteroids (or on physiologic replacement doses only) and stable or improved clinically.
  * PR: Requires:• ≥ 50% decrease compared with baseline in the sum of products of perpendicular diameters of all measurable enhancing lesions sustained for at least 4 weeks. • No progression of nonmeasurable disease. • Stable or improved nonenhancing (T2/FLAIR) lesions on same or lower dose of corticosteroids compared with baseline scan; the corticosteroid dose at the time of the scan evaluation should be no greater than the dose at time of baseline scan. • Stable or improved clinically
Time Frame: Completion of treatment (estimated to be 6 months)
Population: There were not any participants enrolled in Cohort B or Cohort C.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Non-small Cell Lung Cancer w/o Corticosteroids | Cohort B: Epithelial Origin Solid Tumors w/o Corticosteroids | Cohort C: NSCLC or Non-NSCLC w/Corticosteroids
Number analyzed (Participants) | 4 | 0 | 0
Participants | 0 |  |

2. Secondary Outcome: Safety of MEDI4736 in Advanced Solid Epithelial-derived Tumor Patients With Brain Metastases as Measured by Number of Participants With Treatment-emergent Adverse Events
Description: -The severity of AEs will be graded by the investigator according to the CTCAE, Version 4.03
Time Frame: 30 days after completion of treatment (estimated to be 7 months)
Population: There were not any participants enrolled in Cohort B or Cohort C.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Non-small Cell Lung Cancer w/o Corticosteroids | Cohort B: Epithelial Origin Solid Tumors w/o Corticosteroids | Cohort C: NSCLC or Non-NSCLC w/Corticosteroids
Number analyzed (Participants) | 4 | 0 | 0
Participants
  Grade 1 anemia | 1 |  |
  Grade 2 anemia | 1 |  |
  Grade 1 bloating | 1 |  |
  Grade 2 constipation | 1 |  |
  Grade 2 diarrhea | 1 |  |
  Grade 1 nausea | 1 |  |
  Grade 1 chills | 1 |  |
  Grade 2 fever | 1 |  |
  Grade 1 non-cardiac chest pain | 1 |  |
  Grade 1 night sweats | 1 |  |
  Grade 2 sinusitis | 1 |  |
  Grade 1 lymphocyte count decreased | 1 |  |
  Grade 2 lymphocyte count decreased | 2 |  |
  Grade 2 weight loss | 1 |  |
  Grade 1 hypercalcemia | 1 |  |
  Grade 3 hypercalcemia | 1 |  |
  Grade 1 hyponatremia | 1 |  |
  Grade 1 arthralgia | 1 |  |
  Grade 3 paresthesia | 1 |  |
  Grade 1 productive cough | 1 |  |
  Grade 2 post nasal drip | 1 |  |
  Grade 1 hyperhidrosis | 1 |  |
  Grade 1 pruritus | 1 |  |
  Grade 1 hypertension | 1 |  |

3. Secondary Outcome: Overall Disease Control Rate of Intracranial Disease
Description: * Defined as the percentage of patients who achieve a complete response, partial response, or stable disease based on assessment of brain lesions
  * CR: Requires: complete disappearance of all enhancing measurable and nonmeasurable disease sustained for at least 4 weeks; No new lesions; stable or improved nonenhancing (T2/FLAIR) lesions.; off corticosteroids (or on physiologic replacement doses only) and stable or improved clinically.
  * PR: Requires:• ≥ 50% decrease compared with baseline in the sum of products of perpendicular diameters of all measurable enhancing lesions sustained for at least 4 weeks. • No progression of nonmeasurable disease. • Stable or improved nonenhancing (T2/FLAIR) lesions on same or lower dose of corticosteroids compared with baseline scan; the corticosteroid dose at the time of the scan evaluation should be no greater than the dose at time of baseline scan. • Stable or improved clinically
Time Frame: Completion of treatment (estimated to be 6 months)
Population: There were not any participants enrolled in Cohort B or Cohort C.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Non-small Cell Lung Cancer w/o Corticosteroids | Cohort B: Epithelial Origin Solid Tumors w/o Corticosteroids | Cohort C: NSCLC or Non-NSCLC w/Corticosteroids
Number analyzed (Participants) | 4 | 0 | 0
Participants | 2 |  |

4. Secondary Outcome: Overall Response Rate of Extracranial Disease
Description: * Defined as the percentage of patients who achieve a complete response or partial response based on assessment of systemic lesions
  * Complete response: Disappearance of all target lesions, non-target lesions, and normalization of tumor marker level. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  * Partial response: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters
Time Frame: Completion of treatment (estimated to be 6 months)
Population: Two participants were not evaluable in Cohort A as the extracranial response per RECIST was not done. There were not any participants enrolled in Cohort B or Cohort C.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Non-small Cell Lung Cancer w/o Corticosteroids | Cohort B: Epithelial Origin Solid Tumors w/o Corticosteroids | Cohort C: NSCLC or Non-NSCLC w/Corticosteroids
Number analyzed (Participants) | 2 | 0 | 0
Participants | 0 |  |

5. Secondary Outcome: Overall Disease Control Rate of Extracranial Disease
Description: * Defined as the percentage of patients who achieve a complete response, partial response, or stable disease based on assessment of systemic lesions
  * Complete response: Disappearance of all target lesions, non-target lesions, and normalization of tumor marker level. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  * Partial response: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters
  * Stable disease: Neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study
Time Frame: Completion of treatment (estimated to be 6 months)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Non-small Cell Lung Cancer w/o Corticosteroids | Cohort B: Epithelial Origin Solid Tumors w/o Corticosteroids | Cohort C: NSCLC or Non-NSCLC w/Corticosteroids
Number analyzed (Participants) | 2 | 0 | 0
Participants | 1 |  |

6. Secondary Outcome: Overall Response Rate Considering Both Intracranial and Extracranial Disease
Description: * Defined as the percentage of patients who achieve a complete response or partial response based on assessment of brain and systemic lesions
  * Intracranial disease
    * Complete response: Disappearance of all target lesions, non-target lesions, and normalization of tumor marker level. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
    * Partial response: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters
  * Extracranial disease
    * Complete response: Disappearance of all target lesions, non-target lesions, and normalization of tumor marker level. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
    * Partial response: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters
Time Frame: Completion of treatment (estimated to be 6 months)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Non-small Cell Lung Cancer w/o Corticosteroids | Cohort B: Epithelial Origin Solid Tumors w/o Corticosteroids | Cohort C: NSCLC or Non-NSCLC w/Corticosteroids
Number analyzed (Participants) | 2 | 0 | 0
Participants | 0 |  |

7. Secondary Outcome: Overall Disease Control Rate Considering Both Intracranial and Extracranial Disease
Description: * Defined as the percentage of subjects who achieve a complete response, partial response, or stable disease based on assessment of brain and systemic lesions
  * Intracranial disease: response and progression will be evaluated using the updated response assessment criteria for high-grade gliomas: Response Assessment in Neuro-Oncology (RANO) working group guideline
  * Extracranial disease: response and progression will be evaluated using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1)
Time Frame: Completion of treatment (estimated to be 6 months)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Non-small Cell Lung Cancer w/o Corticosteroids | Cohort B: Epithelial Origin Solid Tumors w/o Corticosteroids | Cohort C: NSCLC or Non-NSCLC w/Corticosteroids
Number analyzed (Participants) | 2 | 0 | 0
Participants | 1 |  |

8. Secondary Outcome: Duration of Response of Intracranial Disease
Description: * Defined as the interval from the first documentation of objective response (complete response or partial response) to the earlier of the first documentation of disease progression or death from any cause
  * Intracranial disease: response and progression will be evaluated using the updated response assessment criteria for high-grade gliomas: Response Assessment in Neuro-Oncology (RANO) working group guideline
Time Frame: Completion of treatment (estimated to be 6 months)
Population: None of the participants in Cohort A were evaluable for this outcome measure as they did not have an objective response per RANO guidelines. There were not any participants enrolled to Cohort B or Cohort C.
Arm/Group | Cohort A: Non-small Cell Lung Cancer w/o Corticosteroids | Cohort B: Epithelial Origin Solid Tumors w/o Corticosteroids | Cohort C: NSCLC or Non-NSCLC w/Corticosteroids
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Duration of Response of Extracranial Disease
Description: * Defined as the interval from the first documentation of objective response (complete response or partial response) to the earlier of the first documentation of disease progression or death from any cause
  * Extracranial disease: response and progression will be evaluated using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1)
Time Frame: Completion of treatment (estimated to be 6 months)
Population: Two participants were not evaluable in Cohort A as the extracranial response per RECIST was not done. The remaining two participants were not evaluable for this outcome measure because they didn't have an objective response per RECIST. There were not any participants enrolled in Cohort B or Cohort C.
Arm/Group | Cohort A: Non-small Cell Lung Cancer w/o Corticosteroids | Cohort B: Epithelial Origin Solid Tumors w/o Corticosteroids | Cohort C: NSCLC or Non-NSCLC w/Corticosteroids
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Duration of Response Considering Both Intracranial and Extracranial Disease
Description: * Defined as the interval from the first documentation of objective response (complete response or partial response) to the earlier of the first documentation of disease progression or death from any cause
  * Intracranial disease: response and progression will be evaluated using the updated response assessment criteria for high-grade gliomas: Response Assessment in Neuro-Oncology (RANO) working group guideline
  * Extracranial disease: response and progression will be evaluated using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1)
Time Frame: Completion of treatment (estimated to be 6 months)
Population: Two participants were not evaluable in Cohort A as the extracranial response per RECIST was not done. The remaining two participants were not evaluable for this outcome measure because they didn't have an objective response. There were not any participants enrolled in Cohort B or Cohort C.
Arm/Group | Cohort A: Non-small Cell Lung Cancer w/o Corticosteroids | Cohort B: Epithelial Origin Solid Tumors w/o Corticosteroids | Cohort C: NSCLC or Non-NSCLC w/Corticosteroids
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Progression-free Survival (PFS)
Description: * PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
  * At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression). Unequivocal progression of existing non-target lesions.
Time Frame: Up to 2 years after completion of treatment (estimated to be 2 years and 6 months)
Population: There were not any participants enrolled in Cohort B or Cohort C.
Measure: Median (Full Range); unit: days
Arm/Group | Cohort A: Non-small Cell Lung Cancer w/o Corticosteroids | Cohort B: Epithelial Origin Solid Tumors w/o Corticosteroids | Cohort C: NSCLC or Non-NSCLC w/Corticosteroids
Number analyzed (Participants) | 4 | 0 | 0
days | 51.5 [18 to 64] |  |

12. Secondary Outcome: Overall Survival (OS)
Description: -Defined as the interval from the start of study therapy to death from any cause
Time Frame: Up to 2 years after completion of treatment (estimated to be 2 years and 6 months)
Population: One participant in Cohort A was lost to follow-up and is not evaluable for this outcome measure. There were not any participants enrolled to Cohort B or Cohort C.
Measure: Median (Full Range); unit: days
Arm/Group | Cohort A: Non-small Cell Lung Cancer w/o Corticosteroids | Cohort B: Epithelial Origin Solid Tumors w/o Corticosteroids | Cohort C: NSCLC or Non-NSCLC w/Corticosteroids
Number analyzed (Participants) | 3 | 0 | 0
days | 197 [130 to 262] |  |

ADVERSE EVENTS:
Time Frame: Adverse events were collected starting at baseline and ending 30 days after the completion of treatment.
Description: There were no participants enrolled in Cohort B or C and that is why the number of participants at risk for All-Cause Mortality, Serious Adverse Events, and Other Adverse Events is zero.
Arm/Group | Cohort A: Non-small Cell Lung Cancer w/o Corticosteroids | Cohort B: Epithelial Origin Solid Tumors w/o Corticosteroids | Cohort C: NSCLC or Non-NSCLC w/Corticosteroids
All-Cause Mortality (participants affected / at risk) | 2/4 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 4/4 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Non-small Cell Lung Cancer w/o Corticosteroids (N=4) | Cohort B: Epithelial Origin Solid Tumors w/o Corticosteroids (N=0) | Cohort C: NSCLC or Non-NSCLC w/Corticosteroids (N=0)
Parasthesia (Nervous system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Non-small Cell Lung Cancer w/o Corticosteroids (N=4) | Cohort B: Epithelial Origin Solid Tumors w/o Corticosteroids (N=0) | Cohort C: NSCLC or Non-NSCLC w/Corticosteroids (N=0)
Anemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Bloating (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Chills (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Night sweats (General disorders) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 3 | 0 | 0
Weight loss (Investigations) | 1 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Post nasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-23): https://cdn.clinicaltrials.gov/large-docs/14/NCT02669914/Prot_SAP_000.pdf